CLINICAL TRIAL: NCT01786070
Title: Effect of Nebulized Budesonide on Preventing Postextubation Complications in Critically Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Saeed Abbasi, Assistant Professor in Anesthesiology, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 390104
Record Dates: First submitted 2013-02-02; First posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Respiratory Sounds
MeSH Terms: conditions — Respiratory Sounds | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Budesonide (Active Comparator): Budesonide : 1 mg/4ml every 12 hrs for 48 hrs
  Interventions: Drug: Budesonide
- Placebo (Placebo Comparator): Normal saline at an equivalent volume (4 ml every 12 hrs for 48 hrs)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Budesonide
  Arms: Budesonide
Drug: placebo
  Arms: Placebo

SUMMARY:
The aim of this study is evaluation of the effect of administration nebulized budesonide after extubation. The specific objectives of our study are to determine whether multiple doses of nebulized budesonide are effective to reduce or prevent postextubation edema.

In this double-blind randomized clinical trial study, 70 patients (age between 18 to 65) who are intubated (at least for 48 hours) and now are ready for extubation will be enrolled in the study after obtaining a written informed consent from their parents or guardians.

The investigators divide our patients randomly into two equal groups.

-Patients who are in budesonide group will receive nebulized budesonide (1 mg-every 12 hours; n=35) and patients in placebo group receive placebo (normal saline; n=35) until 48 hours after extubation. If patient have extubation criteria the investigators will extubate him and for 24 hours after, another anesthesiologist who is unaware about kind of medication, will evaluate the patients for severity of stridor. We will record the vital sings and grade of stridor every 6 hour. Respiratory rate (RR), heart rate (HR), blood pressure (BP) and oxygen saturation (SPO2) were recorded for each patient immediately before aerosol administration (time 0) and at 30 and 60 min; and 2,4,8,12,24,36 and 48 hrs. After extubation then the presence of stridor (heard with the aid of stethoscope) was recorded within 48 hr of extubation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients' age 18-55 years old
2. Intubated for more than 48 hours after surgery
3. Met the weaning criteria defined as respiratory rate < 30 breaths / min, negative tidal volume > 5 ml/kg ideal body weight, and shallow index (respiratory rate/tidal volume) < 105 breaths / min/L

Exclusion Criteria:

1. Any history of corticosteroid therapy in previous week
2. Nasal or throat disease / surgery
3. Pulmonary airway disease
4. Gastrointestinal bleeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
post extubation stridor | After extubation until 48 hours
  Until 48 hours after extubation we documented if there is stridor in examination

CONTACTS AND LOCATIONS:
Locations (1):
- Alzahra University Hospital, Isfahan, Isfahan, Iran